CLINICAL TRIAL: NCT03210740
Title: A Phase 2, Single-Center, Randomized, Double- Blind, Parallel-Group, Vehicle-Controlled Study Evaluating the Efficacy and Safety of AM001 Cream in the Treatment of Actinic Keratosis (AK) Lesions
Brief Title: Safety and Efficacy Study of AM001 Cream in the Treatment of Actinic Keratosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AmDerma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AD-AM001-AK1
Record Dates: First submitted 2017-07-05; First posted 2017-07-07 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2018-09

CONDITIONS: Actinic Keratosis
MeSH Terms: conditions — Keratosis, Actinic | interventions — potassium dobesilate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AM001 Cream, 7.5% (Experimental): A white to off-white Cream free from any foreign particles
  Interventions: Drug: AM001 Cream, 7.5%
- Vehicle Cream (Placebo Comparator): A white to off-white Cream free from any foreign particles
  Interventions: Drug: Vehicle Cream

INTERVENTIONS:
Drug: AM001 Cream, 7.5% — Active Cream
  Other Names: Potassium Dobesilate
  Arms: AM001 Cream, 7.5%
Drug: Vehicle Cream — Placeo
  Other Names: Placebo Cream
  Arms: Vehicle Cream

SUMMARY:
To compare the safety and efficacy profiles of AM001 Cream, 7.5% and its vehicle cream in the treatment of Actinic Keratosis (AK) Lesions

DETAILED DESCRIPTION:
A Phase 2, Single-Center, Randomized, Double- Blind, Parallel-Group, Vehicle-Controlled Study Evaluating the Efficacy and Safety of AM001 Cream in the Treatment of Actinic Keratosis (AK) Lesions

ELIGIBILITY:
Inclusion Criteria:

1. Subject must provide written informed consent.
2. Subject must be male or non-pregnant females of any race, and any skin type aged 18 to 80 years both inclusive.
3. Subject has 4 to 8 clinically typical, visible, discrete, nonhyperkeratotic, nonhypertrophic AK lesions, each at least 4 mm in diameter within a 25cm² contiguous treatment area on the face or the balding scalp.
4. Subject is willing to avoid exposure to sunlight, use of tanning booths, sunlamps, or nonprescription UV (ultra-violate) light sources during the study period.ooths, sunlamps, or nonprescription UV (ultra-violate) light sources during the study period.
5. If female subject of childbearing potential, the subject must have a negative urine pregnancy test at Visit 1/ Screening and must have been using an acceptable form of birth control for at least 2 months prior to Visit 1/ Screening and is willing to continue birth control during the study.
6. Subject must be willing and able to understand and comply with the requirements of the study, apply the assigned investigational product as instructed, return for the required study visits, comply with therapy prohibitions.
7. Subject must be in good health, as confirmed by medical history and physical exam, and free from any clinically significant disease/condition, other than actinic keratosis, that might interfere with the study evaluations.

Exclusion Criteria:

1. Subject has very thick and/or hyperkeratotic actinic keratosis AK lesions in the treatment area.
2. Subject has used topical treatment of actinic keratosis in the treatment area with 5-fluorouracil, imiquimod, diclofenac, corticosteroids or retinoids within 1 month prior to Visit 2/Baseline or during the study.
3. Subject has used treatment with PDT (photodynamic therapy) or physical therapies (e. g. cryotherapy, curettage or surgical treatment) in the treatment area within 1 month prior to Visit 2/Baseline or during the study.
4. Subject has used chemical peel, dermabrasion, laser abrasion, PUVA (prosalen plus ultraviolet A) therapy or UVB therapy within 6 months prior to Visit 2/Baseline or during the study.
5. Subject has used immunomodulators or immunosuppressive therapies, interferon, oral corticosteroids, oral retinoids or cytotoxic drugs within 1 month prior to Visit 2/Baseline or during the study.
6. Subject has untreated basal cell carcinoma, squamous cell carcinoma or melanoma in the treatment area.
7. Subject has suntan or tattoos that may interfere with the assessments in the treatment area.
8. Subject has dermatological diseases in the treatment area that may interfere with the assessments, e.g. acute skin inflammation, atopic dermatitis, eczema, rosacea, psoriasis, seborrheic dermatitis, peri-oral dermatitis or hyperpigmentation.
9. Subject who consumes excessive amount of alcohol, abuse or have any condition that in the investigator's opinion would compromise compliance, with this protocol.
10. Subject has history of malignancy not in remission for at least 5 years excluding basal cell carcinoma and nonperiorificial squamous cell carcinoma of the skin.
11. Female subject who is pregnant, nursing or planning a pregnancy within the study participation period
12. Subject has symptoms of a clinically significant illness that may influence the outcome of the study in the 4 weeks prior to Visit 1/Screening.
13. Subject has participated in another clinical trial involving investigational product or device in the 4 weeks prior to Visit 1/Screening.
14. Subject has known allergic reactions to components of the investigational product.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2018-02-13 (Actual); Study Completion 2018-04-24 (Actual)

PRIMARY OUTCOMES:
Complete clearance of all lesions | 8 weeks post treatment
  (100 % of all AK lesions cleared) 8 weeks post treatment

SECONDARY OUTCOMES:
Complete clearance of all baseline lesions weeks of treatment | 16 weeks
  (100% of baseline AK lesions cleared) after 16 weeks of treatment
Complete clearance of all lesions | 12 weeks
  (100% of baseline AK lesions cleared) after 12 weeks of treatment
Complete clearance of all lesions | 8 weeks
  (100% of baseline AK lesions cleared) after 8 weeks of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- AmDerma Pharmaceuticals, LLC, High Point, North Carolina, United States